CLINICAL TRIAL: NCT00540670
Title: A Double-Blind Study of E5555 in Japanese Subjects With Coronary Artery Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E5555-J081-206
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2010-02

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — E 5555

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: E5555 50 mg
- 2 (Experimental)
  Interventions: Drug: E5555 100 mg
- 3 (Experimental)
  Interventions: Drug: E5555 200 mg
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E5555 50 mg — E5555 50 mg (tablet) taken orally, once a day.
  Arms: 1
Drug: E5555 100 mg — E5555 100 mg (tablet) taken orally, once a day.
  Arms: 2
Drug: E5555 200 mg — E5555 200 mg (tablet) taken orally, once a day.
  Arms: 3
Drug: Placebo — Placebo (tablet) taken orally, once a day.
  Arms: 4

SUMMARY:
The purpose of this study is to assess the safety and tolerability of E5555 in Japanese subjects with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

1. 45 - 80 years old (at time of informed consent).
2. Male or female (females of childbearing potential must use contraception).
3. Confirmed coronary artery disease.
4. All subjects must be receiving aspirin (75 - 325 mg).

Exclusion Criteria:

1. Unwilling or unable to provide informed consent.
2. History of acquired or congenital bleeding disorder, coagulopathy, or platelet disorder.
3. Recent trauma or major surgery.
4. Evidence of active pathological bleeding or history of bleeding such as gastrointestinal or genitourinary, unless the cause has been definitely corrected.
5. History of intracranial bleeding or history of hemorrhagic retinopathy.
6. New York Heart Association class III or IV congestive heart failure.
7. Pregnant or lactating women.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Adverse events, bleeding events, clinical laboratory tests, Coagulation tests, vital signs and 12-lead ECG | 6 months

SECONDARY OUTCOMES:
Major cardiac adverse events, biomarkers, platelet aggregation inhibition, plasma concentration. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Masaru Takeuchi, Study Director — New Product Development, Clinical Research Center, Eisai Co., Ltd.
Locations (25):
- Japan (25):
  - Ichinomiya, Aichi-ken
  - Gifu, Gifu
  - Ōgaki, Gifu
  - Asahikawa, Hokkaido
  - Chitose, Hokkaido
  - Sapporo, Hokkaido
  - Tomakomai, Hokkaido
  - Himeji, Hyōgo
  - Nishinomiya, Hyōgo
  - Tsuchiura, Ibaraki
  - Kanazawa, Ishikawa-ken
  - Yokohama, Kanagawa
  - Kumamoto, Kumamoto
  - Matsusaka, Mie-ken
  - Tsu, Mie-ken
  - Osaka, Osaka
  - Sayama, Osaka
  - Kitamoto, Saitama
  - Saitama, Saitama
  - Shizuoka, Shizuoka
  - Bunkyo-ku, Tokyo
  - Musashino, Tokyo
  - Ōta-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Tachikawa, Tokyo